CLINICAL TRIAL: NCT01699347
Title: Cohort Prospective Study of Children With Head and Neck Cystic Malformation Who Are Treated With Intracystic OK432
Acronym: OK432
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Carmel Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CMC-11-0059-CTIL
Record Dates: First submitted 2012-08-19; First posted 2012-10-03 (Estimated); Last update posted 2013-12-02 (Estimated); Status verified 2013-11

CONDITIONS: CYSTIC MALFORMATION
Keywords: OK432, CYSTIC MALFORMATION
MeSH Terms: interventions — Picibanil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- OK432 (Experimental): Intracystic injection of OK432 under US guiding
  Interventions: Drug: Intracystic injection of OK432 under US guiding

INTERVENTIONS:
Drug: Intracystic injection of OK432 under US guiding — Intracystic injection of OK432 under US guiding
  Other Names: OK432 (Picibanil)

SUMMARY:
Cohort study evaluate the efficacy treatment with OK-432 in cystic malformation of the head and neck region.

The malformations are macrocystic and the preevaluation will include CT/MRI, US and blood tests.

The injection will be in the OR under US guided, maximal dose will be 0.2mg. The follow-up will be of short term - till 30 days post injection and long term - follow-up wil be till 2 years.

DETAILED DESCRIPTION:
A cohort study, before the injection all the patients in the study will go through:

1. CT/MRI
2. US to estimate the cyst size
3. CBC, PT, PTT, INR, ASLO
4. ECG If the patient is qualified to the study the parent will sign on the inform consent, than the child will be photographed AP and lateral.

The injection will be held in the OR under US guidance with 18q20 gauge needle, first all the cyst contents will be sucked than the OK432 will be injected in.

After the injection the child will stay for one night if it was general anesthesia and 4 hours in the case of local anesthesia.

Short term follow - 3-5 days with the phone, up: till 30 days from the injection with US, stills photo.

Long term follow-up: 6 months, 1 year, 2 years

ELIGIBILITY:
Inclusion Criteria:

* LYMPHATIC MALFORMATION MACROCYSTIC OR MIXED WITH MORE THEN 50% MACROCYSTIC.
* ONLY IN THE HEAD AND NECK AREA
* TIME FROM OPERATION AT LEAST 6 MONTHS

Exclusion Criteria:

* penicillin allergy
* pregnancy
* familial history of RF
* Post streptococcal glomerulonephritis
* Background illness-heart, kidney, lungs
* fever > 38.5c in the op day
* URT Infection
* Family history of PANDAS

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 5 (Estimated)
Dates: Start 2012-09; Primary Completion 2014-01 (Estimated); Study Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
evaluation of the efficacy in treating cystic malformation with OK432 by measuring time that elapsed without recurrence | 4 years

SECONDARY OUTCOMES:
TREATMENT SAFETY BY no. of participants with adverse events | 4 YEARS

CONTACTS AND LOCATIONS:
Overall Officials: Raanan Cohen-Kerem, MD, Principal Investigator — Carmel Medical Center, Haifa, Israel
Locations (1):
- Department of Otolaryngology, Carmel Medical Center, Haifa, Israel